CLINICAL TRIAL: NCT02021214
Title: Effects of Methylphenidate (Ritalin®) on the Neural Basis of Anxiety: a Placebo-controlled fMRI Study in Healthy Male Subjects
Brief Title: Effects of Methylphenidate (Ritalin®) on the Neural Basis of Anxiety
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 131297
Record Dates: First submitted 2013-12-09; First posted 2013-12-27 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: PTSD
Keywords: Methylphenidate; Fear extinction; fMRI; mPFC
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Double-blind, cross-over design with two drug conditions. Drug conditions are placebo and methylphenidate 40 mg. Order will be balanced and pseudo-random.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylphenidate/Placebo (Experimental): 40 mg Methylphenidate, per os, single dose Placebo, single dose
  Interventions: Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate
  Other Names: Ritalin
Drug: Placebo

SUMMARY:
In the present study, investigator will investigate the effects of methylphenidate (40 mg) on mPFC activity in healthy male volunteers during fear extinction using functional magnetic resonance imaging (fMRI). Additionally, investigators will examine the effects of methylphenidate during aversive interoceptve arousal. The present study will help to identify brain structures and networks involved in anxiety and will give insights for methylphenidate as a possible adjunct to behavioral therapy for patients with anxiety disorders. Further, this study may provide important information about the possible use of fMRI to help the development of drugs for the treatment of anxiety disorders.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) affects 5-10% of the general U.S. population at some point during their lifetime; however, the prevalence in much higher among certain subgroups, including active duty military personnel and veterans. Pharmacotherapy of PTSD has made little headway on the past two decades. Methylphenidate (Ritalin®) is a stimulant drug that amplifies dopaminergic and noradrenergic signaling in the brain. Dopamine and norepinephrine are thought to play a critical role during fear extinction by moderating medial prefrontal cortex (mPFC) activity. The magnitude of mPFC activity seems to crucially affect the degree of fear extinction. The model of fear extinction is one approach to conceptualize PTSD. Thereby a previously neutral stimulus is paired with a highly aversive unconditioned stimulus. Fear extinction refers to the decrement in that conditioned fear responses that occur with repeated presentation of the conditioned neutral fear stimulus without the aversive stimulus. While preclinical data suggest that a single dose of methylphenidate enhances fear extinction, it is less clear how methylphenidate affects fear extinction in humans. However, exposing PTSD patients to new therapies is difficult. In the present study, investigator will investigate the effects of methylphenidate (40 mg) on mPFC activity in healthy male volunteers during fear extinction using functional magnetic resonance imaging (fMRI). Additionally, investigators will examine the effects of methylphenidate during aversive interoceptve arousal. The present study will help to identify brain structures and networks involved in anxiety and will give insights for methylphenidate as a possible adjunct to behavioral therapy for patients with anxiety disorders. Further, this study may provide important information about the possible use of fMRI to help the development of drugs for the treatment of anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 to 40 years of age, inclusive.
* In good general health (as determined by medical history, blood pressure, and ECG), especially no findings (including concomitant medications) that would constitute contraindications for treatment with any of the study drugs.
* A weight of > 120 lbs (55 kg) and a BMI between 18 to 30 kg/m2, inclusive.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) the day before and during the study day.
* Subjects able to participate and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular (including structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease or myocardial infarction), renal or CNS disease (including seizures), gallbladder removal or other medical or surgical condition that could alter the absorption, metabolism or elimination of drugs.
* Family history of sudden death or ventricular arrhythmia.
* Any major illness (as judged by the study physician) within 1 month prior to first dose.
* Current or history of any psychiatric disorder, marked anxiety, tension and agitation.
* History of glaucoma.
* History (including family history) of motor tic or diagnosis of Tourette's syndrome.
* History of psychotropic medicine and/or alcohol dependence.
* Active suicidal ideation, history of suicidal behavior, or otherwise considered at high suicidal risk by trained study staff using the C-SSRS.
* Positive urine toxicology (drugs of abuse as determined by a positive urine test) at screening and before each drug administration.
* Use of any medications or herbal remedies, including psychotropic medicines and regular sleep medications, taken within 14 days or 6 times the elimination half-life of the medication (whichever is longer) prior to the first dose and throughout the study, with the exception of acetaminophen for minor pains, occasional use of sleeping medication as long as it is not taken the evening prior to a visit, medications explicitly approved by the investigator and the sponsor.
* Past intolerance (including allergic) to any of the study medications or components thereof.
* Supine systolic blood pressure (BP) >140 or >90 mmHg, diastolic BP <90 mmHg or <50 mmHg (mean of two measurements at screening) and current or past history of clinically significant hypertension.
* Current smoker (> 10 cigarettes/day); habitual caffeine consumption of more than 400 mg/d (approximately 4 cups of coffee or equivalent).
* QTcF > 450 msec based on the average interval on triplicate ECGs. Notable resting bradycardia (mean HR < 45 bpm) or notable resting tachycardia (mean HR > 90 bpm).
* Contraindication to magnetic resonance imaging.
* Participation in a clinical trial with an investigational drug or a device within 30 days prior to dosing in the first period.
* Volunteers who do not have sufficient command of the English language, or who have any other impairment that would prevent them from reading and understanding the informed consent form(s) and completing the study procedures including clinical testing.
* Any other reason why, per study physician, the subject should not participate in this study, including concomitant disease or condition that could interfere with, or for which the study drug might interfere with, the conduct of the study, or that would, in the opinion of the principal investigator, pose an unacceptable risk to the subject in this study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in blood oxygenation level-dependent BOLD signal responses | 6 hours
  Methylphenidate-induced changes in BOLD signal responses in brain regions relevant in fear disorders (e.g. amygdala, insula, and prefrontal cortex) during a fear extinction task compared to placebo.

SECONDARY OUTCOMES:
Changes in BOLD signal responses | 6 hours
  Methylphenidate induced changes in BOLD signal responses in regions implicated in emotional processing while anticipating a positive interoceptive stimulus compared to placebo.
Changes in skin conductance response | 6 hours
  Changes compared to placebo in skin conductance respo during a fear extinction task
Latency and accuracy during a interoceptive stimulus task | 2 hours
  This task aims to examine the participants' response to an aversive interoceptive stimulus. Individuals will perform a simple continuous performance task during the paradigm. Subjects are asked to press one of three buttons to rate the images on the screen as either 'dislike', 'neutral' or 'like'. Both accuracy and response latency (ms) will be recorded to determine effects of anticipation and stimulus presentation

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Paulus, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Psychiatry Clinical Research, San Diego, California, United States